CLINICAL TRIAL: NCT00171808
Title: Phase II Study on Letrozole in Patients With Advanced or Recurrent Hormone Receptor Positive Endometrial Cancer
Brief Title: Letrozole in the Treatment of Advanced or Recurrent Hormone Receptor Positive Endometrial Cancer
Acronym: deFEND
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CFEM345ADE08; EudraCT-Number: 2004-003886-34 (Registry Identifier: EudraCT)
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Endometrial Cancer
Keywords: Endometrial Cancer; Aromatase inhibitor; Advanced or recurrent; hormone receptor positive
MeSH Terms: conditions — Endometrial Neoplasms; Recurrence | interventions — Letrozole

ARMS (1):
- Letrozole (Experimental)
  Interventions: Drug: Letrozole

INTERVENTIONS:
Drug: Letrozole

SUMMARY:
In Western industrialized countries, endometrial cancer is the most common malignancy of the female reproductive tract.

The general therapy options are surgery, radiotherapy, chemotherapy and endocrine therapy. This trial will investigate the efficacy and safety of letrozole in the treatment of advanced or recurrent hormone receptor-positive endometrial cancer .

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age > 18 years
* Presence of histologically proven adenocarcinoma or adenosquamous carcinoma of the endometrium
* Presence of advanced or recurrent endometrial cancer, FIGO stage I-IV, incurable with surgery and/or radiation therapy
* Documented ER and/or PgR positive endometrial cancer. Hormone receptor positivity is defined according to routine practice at each participating laboratory.
* Patient must be postmenopausal defined as

  * Age ≥55 years.
  * Age <55 but no spontaneous menses for at least 1 year.
  * Age <55 and spontaneous menses within the past 1 year, but currently amenorrheic (e.g., spontaneous or secondary to hysterectomy), and with postmenopausal gonadotrophin levels (luteinizing hormone and follicle stimulating hormone levels >40 IU/L) or postmenopausal estradiol levels (<5 ng/dL) or according to the definition of "postmenopausal range" for the laboratory involved.
  * Bilateral oophorectomy
  * Radiation menopause
* Presence of measurable disease (by clinical/radiological examination - according to RECIST criteria : minimum indicator lesion size : 20 mm (unless spiral CT scan in which case > 10 mm)
* ECOG performance status of 0, 1 or 2
* Adequate bone marrow function (WBC ≥ 3.5 x 1'000'000'000/L and platelets ≥ 100.0 x 1'000'000'000/L) and hemoglobin > 10.0 g/dl
* Adequate renal function (creatinine < 120 µmol/L) and hepatic function (bilirubin < 25 µmol/L, AST (SGOT < 60 U/L)
* Minimum life expectancy of at least 6 months
* Patients who are accessible for treatment and follow-up

Exclusion Criteria:

* Presence of non-measurable disease only
* Other concomitant anti-cancer treatment (except external radiation treatment [XRT] for symptomatic metastatic lesions if other assessable untreated lesions are present)
* Prior treatment with aromatase inhibitors or anti-estrogens (up to one previous progestational hormone therapy regimen for recurrent disease is permitted)
* Clear cell or papillary serous histology, uterine sarcomas, mixed Mullerian tumors (MMT) and/or adenosarcomas
* Other concurrent malignant disease with the exception of cone-biopsied in situ carcinoma of the cervix uteri, or adequately treated basal or squamous cell carcinoma of the skin, or other curable cancers e.g. Hodgkin's disease or non-Hodgkin lymphoma (NHL), provided 5 years have elapsed from completion of therapy, and there has been no recurrence
* Known central nervous system (CNS) metastases, bilateral diffuse lymphangiosis carcinoma of the lung (>50 % of lung involvement, or dyspnea at rest requiring supplemental oxygen therapy), evidence of metastases estimated as more than a third of the liver as defined by sonogram and/or CT scan
* Uncontrolled endocrine disorders such as diabetes mellitus, confirmed hypo- or hyperthyroidism, Cushing's Syndrome, Addison's disease (treated or untreated)
* Unstable angina and uncontrolled cardiac disease
* Treatment with other investigational drugs (drugs not marketed for any indication) within the past 30 days and/or the concomitant use of investigational drugs
* A history of non-compliance to medical regimens and patients who, in the opinion of the investigator, are unlikely to cooperate fully during the study
* Inability to swallow pills

Additional protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2005-04; Primary Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
clinical response rate (partial response PR and complete response CR) according to RECIST at least once during the treatment period | until disease progression

SECONDARY OUTCOMES:
Time to progression (TTP) | until disease progression
Overall survival (OS) | until disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmeceuticals
Locations (15):
- Germany (15):
  - Ebersberg, Germany, Celle
  - Heidelberg, Germany, Ebersberg
  - Novartis Investigative Site, Freiburg im Breisgau
  - Ebersberg, Germany, Hamburg
  - Novartis Investigative Site, Hamburg
  - Celle, Germany, Hanover
  - Tuebingen, Germany, Heidelberg
  - Novartis Investigative Site, Karlsruhe
  - Muenchen, Germany, Kiel
  - Muenchen, Germany, München
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Oberaudorf
  - Novartis Investigative Site, Rostock
  - Novartis Investigative Site, Tübingen
  - Hannover, Germany, Wolfsburg

REFERENCES:
- See also: Abstract Page 39 (ISSN 1048891X) — http://journals.lww.com/ijgc/Documents/ESGO%202011%20Abstracts.pdf